CLINICAL TRIAL: NCT04015739
Title: A GINECO Phase II Trialo Assessing the Safety and the Efficacy of the Bevacizumab, Olaparib and Durvalumab (MEDI 4736) Combination in Patients With Advanced Epithelial Ovarian Cancer in Relapse
Brief Title: Tri Association in Patient With Advanced Epithelial Ovarian Cancer in Relapse
Acronym: BOLD
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: ARCAGY/ GINECO GROUP (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GINECO OV 238
Record Dates: First submitted 2019-01-02; First posted 2019-07-11 (Actual); Last update posted 2022-08-17 (Actual); Status verified 2022-08

CONDITIONS: Epithelial Ovarian Cancer; Relapse
Keywords: Bevacizumab; Olaparib; Durvalumab; Tri association
MeSH Terms: conditions — Carcinoma, Ovarian Epithelial; Recurrence | interventions — Bevacizumab; olaparib; durvalumab

STUDY DESIGN:
Intervention Model Description: Patients will be treated the same way in the PRR and PSR cohorts:
  Durvalumab 1.12 g IV on Day 1 Q3W Bevacizumab 15 mg/kg Day 1 Q3W Olaparib 300 mg bid po, continuously
  Patients will be treated upon disease progression, unacceptable toxicity or consent withdrawal.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Bevacizumab, Olaparib and Durvalumab (Experimental): Single arm study
  Interventions: Drug: Bevacizumab, Olaparib and Durvalumab (MEDI 4736) combination

INTERVENTIONS:
Drug: Bevacizumab, Olaparib and Durvalumab (MEDI 4736) combination — Patients will receive a combination of these 3 drugs :
  Bevacizumab 15mg/kg q3w IV, Olaparib 300mg BD Per Os; and Durvalumab (MEDI 4736) 1.12g IV q3w
  Other Names: Experimental treatment

SUMMARY:
Assessing the safety and efficacy of the bevacizumab, Olaparib and Durvalumab (MEDI 4736) combination in patient with high grade serous or high grade endometrioid or other high grade epithelial non mucinous ovarian tumor, with at least one previous line of platinum-taxane chemotherapy, and present with platinum resistant disease (PRR) or platinum-sensitive relapse (PSR), whatever the line of chemotherapy given at relapse.

DETAILED DESCRIPTION:
Bevacizumab and olaparib have already been tested on 12 patients in a phase I trial at their usual doses (10 mg/kg q2w and 400 mg bid - 50 mg capsules -, respectively), and no DLTs were observed. The addition of an anti-VEGF small molecule, cediranib, to olaparib doubled the median PFS in a randomized phase II trial in patients with platinum sensitive relapse, with a manageable safety profile.

A recently reported phase I trial established the RDP2D of Durvalumab and Olaparib - 150 mg tablets -, when given in combination, at 1500 mg every 4 weeks, and 300 mg bid, respectively. In addition, the ENGOT/GINECO PAOLA phase III trial is currently evaluating the combination of Olaparib and Bevacizumab as first-line maintenance after platinum-paclitaxel combination, in patients with advanced high-grade serous ovarian carcinoma. Under the hypothesis of a survival benefit in favor of this combination, it would also be of interest to assess the value of adding Durvalumab in order to improve the efficacy of the overall combination.

There are no trials to date assessing anti-VEGF in combination with anti-PARP and anti-PD-L1 therapy.

Beside additive efficacy, a synergistic effect could be expected :

* Between bevacizumab and durvalumab, through normalization of blood vessel and potentiation of immunologic infiltration.
* Between olaparib and durvalumab, through cytotoxicity-mediated release of antigens and impairment of mutation repair mechanisms, thereby increasing neoantigen loads.
* Between olaparib and bevacizumab, through tumor environment modulation and signaling of DNA damage inhibition, which has already been tested with the anti-VEGF cediranib.

For those reasons the sponsor propose a phase II trial of Olaparib, Bevacizumab and Durvalumab combination, in patients with relapsing AO high grade carcinoma :

* In platinum sensitive relapse (PSR), whatever the line, in patients not amenable to frontline surgery of the relapse and previously-treated by a platinum-containing chemotherapy in first line and

  * Either didn't receive any of the tested drugs,
  * Or previously received either bevacizumab or olaparib BUT NOT the combination of both drugs.
* In platinum-resistant relapse (PRR), in previously untreated patients for their relapse, or in patients who received a maximum of 1 chemotherapy regimen in this setting and either

  * Either didn't receive any of the tested drugs,
  * Or previously received either bevacizumab or olaparib BUT NOT the combination of both drugs.

The trial will also propose translational research, including :

* Assessment of germline and somatic BRCA mutations and determination of HRD phenotype and mutational load by NGS
* Quantification of mutagenesis in simultaneous treatment on ctDNA
* Characterization of immune response in the tumor by Nanostring immuno-oncology panel on tumors

ELIGIBILITY:
Inclusion Criteria:

Patients with platinum resistant relapse

* Female Patient must be ≥18 years of age.
* Signed informed consent and ability to comply with treatment and follow-up.
* Patient with Ovarian cancer, primary peritoneal cancer and/or fallopian-tube cancer, histologically confirmed (based on local histopathological findings): high grade serous or high grade endometrioid or other high grade epithelial non mucinous ovarian tumor.
* Patient who has completed at least one line of platinum-taxane chemotherapy, and presents with platinum resistant relapse (resistant disease defined by a tumor progression less than six months after the last dose of platinum) [Note: the patient may have received one or even more line of platinum based chemotherapy] OR Patient who is in platinum-sensitive relapse, whatever the line of chemotherapy given at relapse [Note: any chemotherapy previously administered must have contained a platinum compound]. The platinum sensitive relapse is defined by a tumor progression occurring more than six months after the last dose of platinum chemotherapy.
* Patient who didn't receive any of the tested drugs, or previously received either bevacizumab or olaparib BUT NOT the combination of both drugs.
* At least one measurable or evaluable lesion that can be accurately assessed at baseline by computed tomography (CT) (or magnetic resonance imaging [MRI] where CT is contraindicated) and is suitable for repeated assessment as per irRC. The baseline scan must be obtained within 28 days of first dose.
* Availability of a pre-treatment tumor sample (archival FFPE block or fresh biopsy if feasible) lasting of less than 3 months before inclusion into the study and performed AFTER the last chemotherapy administration.
* Patient not amenable to cytoreductive surgery at the time of relapse (surgery is not allowed during the protocole treatment).
* Patient must have normal organ and bone marrow function:

  * Hemoglobin ≥ 10.0 g/dL. (Transfusions is not allowed within 28 days before randomization)
  * Absolute neutrophil count (ANC) ≥ 1.5 x 109/L.
  * Platelet count ≥ 100 x 109/L. (Platelet transfusion or G-CSF administration is not allowed within 28 days before randomization)
  * Total bilirubin ≤ 1.5 x institutional upper limit of normal (ULN).
  * Aspartate aminotransferase / Serum Glutamic Oxaloacetic Transaminase (ASAT/SGOT)) and Alanine aminotransferase / Serum Glutamic Pyruvate Transaminase (ALAT/SGPT)) ≤ 2.5 x ULN, unless liver metastases are present in which case they must be ≤ 5 x ULN.
  * Creatinine clearance ≥ 60 mL/min by Cockcroft and Gault formula.
  * Patient not receiving anticoagulant medication who has an International Normalized Ratio (INR) ≤ 1.5 and an Activated ProThrombin Time (aPTT) ≤ 1.5 x ULN. The use of full-dose oral or parenteral anticoagulants is permitted as long as the INR or APTT is within therapeutic limits (according to site medical standard). If the patient is on oral anticoagulants, dose has to be stable for at least two weeks at the time of inclusion.
  * Urine dipstick for proteinuria < 2+. If urine dipstick is ≥ 2+, 24-hour urine must demonstrate < 1 g of protein in 24 hours.
  * Normal blood pressure or adequately treated and controlled hypertension (systolic BP ≤ 150 mmHg and/or diastolic BP ≤ 90 mmHg).
* Expectancy of at least 12 weeks
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1.
* Postmenopausal or evidence of non-childbearing status for women of childbearing potential prior to the first dose of study treatment (see protocol appendix 1).
* As this study will include patients in France, a subject will be eligible for inclusion in this study only if either affiliated to, or a beneficiary of, a social category.

Patients with platinum sensitive relapse

* Female Patient must be ≥18 years of age.
* Signed informed consent and ability to comply with treatment and follow-up.
* Patient with :
* Ovarian cancer, primary peritoneal cancer and/or fallopian-tube cancer, histologically confirmed (based on local histopathological findings): high grade serous or high grade endometrioid or other high grade epithelial non mucinous ovarian tumor.
* Patient who is in platinum-sensitive relapse, whatever the line of chemotherapy given at relapse [Note: any chemotherapy previously administered must have contained a platinum compound]. The platinum sensitive relapse is defined by a tumor progression occurring more than six months after the last dose of platinum chemotherapy.
* Patient who didn't receive any of the tested drugs, or previously received either bevacizumab or olaparib BUT NOT the combination of both drugs.
* At least one measurable or evaluable lesion that can be accurately assessed at baseline by computed tomography (CT) (or magnetic resonance imaging [MRI] where CT is contraindicated) and is suitable for repeated assessment as per irRC. The baseline scan must be obtained within 28 days of first dose.
* Availability of a pre-treatment tumor sample (archival FFPE block or fresh biopsy if feasible) lasting of less than 3 month before inclusion into the study and performed AFTER the last chemotherapy administration.
* Patient not amenable to cytoreductive surgery at the time of relapse (surgery is not allowed during the protocole treatment).
* Patient must have normal organ and bone marrow function:

  * Hemoglobin ≥ 10.0 g/dL. (Transfusions is not allowed within 28 before randomization)
  * Absolute neutrophil count (ANC) ≥ 1.5 x 109/L.
  * Platelet count ≥ 100 x 109/L. (Platelet transfusion or G-CSF administration is not allowed within 28 days before randomization).
  * Total bilirubin ≤ 1.5 x institutional upper limit of normal (ULN).
  * Aspartate aminotransferase / Serum Glutamic Oxaloacetic Transaminase (ASAT/SGOT)) and Alanine aminotransferase / Serum Glutamic Pyruvate Transaminase (ALAT/SGPT)) ≤ 2.5 x ULN, unless liver metastases are present in which case they must be ≤ 5 x ULN.
  * Creatinine clearance ≥ 60 mL/min by Cockcroft and Gault formula.
  * Patient not receiving anticoagulant medication who has an International Normalized Ratio (INR) ≤ 1.5 and an Activated ProThrombin Time (aPTT) ≤ 1.5 x ULN. The use of full-dose oral or parenteral anticoagulants is permitted as long as the INR or APTT is within therapeutic limits (according to site medical standard). If the patient is on oral anticoagulants, dose has to be stable for at least two weeks at the time of incusion.
  * Urine dipstick for proteinuria < 2+. If urine dipstick is ≥ 2+, 24-hour urine must demonstrate < 1 g of protein in 24 hours.
  * Normal blood pressure or adequately treated and controlled hypertension (systolic BP ≤ 150 mmHg and/or diastolic BP ≤ 90 mmHg).
* Expectancy of at least 12 weeks
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1.
* Postmenopausal or evidence of non-childbearing status for women of childbearing potential prior to the first dose of study treatment.
* As this study will include patients in France, a subject will be eligible for inclusion in this study only if either affiliated to, or a beneficiary of, a social category.

Exclusion Criteria:

* Non-epithelial origin of the tumor (i.e. germ cell tumor).
* Ovarian tumors of low malignant potential (e.g. borderline tumors), or mucinous carcinoma.
* Carcinosarcoma (Mixed Mullerian Tumor)
* Patient with synchronous primary endometrial cancer unless both of the following criteria are met:

  * Stage < II,
  * Less than 60 years old at the time of diagnosis of endometrial cancer with stage IA or IB grade 1 or 2, or stage IA grade III endometrial carcinoma,OR ≥ 60 years old at the time of diagnosis of endometrial cancer with stage IA grade 1 or 2 endometrioid adenocarcinoma.

Patient with serous or clear cell adenocarcinoma or carcinosarcoma of the endometrium is not eligible.

* Other malignancy within the last 5 years except: adequately treated non-melanoma skin cancer, curatively treated in situ cancer of the cervix, ductal carcinoma in situ (DCIS). Patient with a history of localized malignancy diagnosed over 5 years ago may be eligible provided she completed her adjuvant systemic therapy and remains free of recurrent or metastatic disease. Patient with history of primary triple negative breast cancer may be eligible provided she completed her definitive anticancer treatment more than 3 years ago and she remains breast cancer disease free prior to start of study treatment.
* Patient with myelodysplastic syndrome/acute myeloid leukemia history.
* Current or prior use of immunosuppressive medication within 14 days (use 28 days if combining durvalumab with a novel agent) before the first dose of durvalumab, with the exceptions of intranasal and inhaled corticosteroids or systemic corticosteroids at physiological doses, which are not to exceed 10 mg/day of prednisone, or an equivalent corticosteroid. (...)
* Any unresolved toxicity NCI CTCAE Grade ≥2 from previous anticancer therapy with the exception of alopecia, vitiligo, and the laboratory values defined in the inclusion criteria

  * Patients with Grade ≥2 neuropathy will be evaluated on a case-by-case basis after consultation with the Study Physician.
  * Patients with irreversible toxicity not reasonably expected to be exacerbated by treatment with durvalumab may be included only after consultation with the Study Physician.
* Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease [e.g., colitis or Crohn's disease], diverticulitis [with the exception of diverticulosis], systemic lupus erythematosus, Sarcoidosis syndrome, or Wegener syndrome [granulomatosis with polyangiitis, Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, etc]). (...)
* Patient receiving radiotherapy within 6 weeks prior to study treatment.
* Major surgery within 4 weeks of starting study treatment and patient must have recovered from any effects of any major surgery.
* Previous allogenic bone marrow transplant.
* Any previous treatment with Anti PD(L)-1 immunotherapy, including durvalumab
* Any previous treatment with a PARP inhibitor in combination with an anti-VEGF (previous treatment with PARP inhibitor alone or anti-VEGF alone is allowed).
* Past medical history of interstitial lung disease, drug-induced pneumonitis, radiation pneumonitis that required steroid treatment, or any evidence of clinically active interstitial lung disease
* Administration of other simultaneous chemotherapy drugs, any other anticancer therapy or anti-neoplastic hormonal therapy, or simultaneous radiotherapy during the trial treatment period (hormonal replacement therapy is permitted as are steroidal antiemetics).
* Current or recent (within 10 days prior to inclusion) chronic use of aspirin > 325 mg/day.
* Concomitant use of known potent CYP3A4 inhibitors such as ketoconazole, itraconazole, ritonavir, indinavir, saquinavir, telithromycin, clarithromycin and nelfinavir. The required washout period prior to starting study treatment is 2 weeks.
* Concomitant use of known strong (e.g. phenobarbital, enzalutamide, phenytoin, rifampicin, rifabutin, rifapentine, carbamazepine, nevirapine and St John's Wort) or moderate CYP3A inducers (e.g. bosentan, efavirenz, modafinil). The required washout period prior to starting study treatment is 5 weeks for enzalutamide or phenobarbital and 3 weeks for other agents. Patients should stop using herbal remedies 7 days prior to the first dose of study medication and for the duration of the trial.
* Prior history of hypertensive crisis (CTC-AE grade 4) or hypertensive encephalopathy.
* Clinically significant (e.g. active) cardiovascular disease, Previous Cerebro-Vascular Accident (CVA), Transient Ischemic Attack (TIA) or Sub- Arachnoids Hemorrhage (SAH) within 6 months prior to inclusion.
* History Clinically significant (e.g. active) cardiovascular disease (...)
* Evidence of bleeding diathesis or significant coagulopathy (in the absence of coagulation).
* History or clinical suspicion of brain metastases or spinal cord compression. CT/MRI of the brain is mandatory (within 4 weeks prior to inclusion) in case of suspected brain metastases. Spinal MRI is mandatory (within 4 weeks prior to inclusion) in case of suspected spinal cord compression.
* Significant traumatic injury during 4 weeks prior to inclusion.
* Non-healing wound, active ulcer or bone fracture. Patient with granulating incisions healing by secondary intention with no evidence of facial dehiscence or infection is eligible but require 3 weekly wound examinations.
* History of VEGF therapy related abdominal fistula or gastrointestinal perforation or active gastrointestinal bleeding within 6 months prior to the first study treatment.
* Current, clinically relevant bowel obstruction, including sub-occlusive and occlusive disease.
* Patient with evidence of abdominal free air not explained by paracentesis or recent surgical procedure.
* Evidence of any other disease, metabolic dysfunction, physical examination finding or laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or puts the patient at high risk for treatment related complications.
* Pregnant or lactating women.
* Participation in another clinical study with an investigational product during her chemotherapy course immediately prior to inclusion.
* Patient unable to swallow orally administered medication and patient with gastrointestinal disorders likely to interfere with absorption of the study medication.
* Patient with a known hypersensitivity to olaparib, durvalumab or bevacizumab or any of the recipients of those products.
* Immunocompromised patient, e.g., with known active hepatitis (i.e. Hepatitis B or C) due to risk of transmitting the infection through blood or other body fluids or patient who is known to be serologically positive for human immunodeficiency virus (HIV).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2024-01-29 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability of the PRR cohort: Rate of clinical and radiological non-progressive disease | At 3 months
  Rate of clinical and radiological non-progressive disease, as assessed by immune-related response criteria (irRC) at 3 months
Safety and tolerability of the PSR cohort: Rate of clinical and radiological non-progressive disease | At 6 months
  Rate of clinical and radiological non-progressive disease, as assessed by immune-related response criteria (irRC) at 6 months

SECONDARY OUTCOMES:
CA 125 change as expressed by the KELIM parameter | up to 60 months
  The CA 125 decline will be calculated between inclusion and end of follow-up. Summarize by mean (SD) or median (25 and 75 percentils) depending if the data distribution is normal or not.
Progression free survival (PFS) | up to 60 months
  The PFS wil be calculated between the date of inclusion and the date of progression or death. The follow-up of patients still alive without progression will be censored at the date of the last follow-up visit. The PFS curves will be estimated using Kaplan-Meier methods
Overall survival (OS) | up to 60 months
  The time to death wil be calculated between the date of inclusion and the date of death. The follow-up of patients still alive will be censored at the date of the last follow-up visit. Data on patients lost to follow-up will censored at the date of the administrative inquiry. The survival curves will be estimated using Kaplan-Meier method.
Tumor response | up to 60 months
  The tumour response will be described using the overall response categories,according irRC criteria. Frequecy and percentages will be calculated by category.
Toxicity as assessed by CTCAE V.5.0 scale | up to 60 months
  Frequency and percentages of patients who had at least one AE will be calculated by category:
  * Any adverse event (AE)
  * Any AE related to study drug
  * Any AE leading to permanent study drug discontinuation
  * Any serious AE
  * Any serious AE related to study drug
  * Any serious AE leading to permanent study drug discontinuation
  When n = 5 for PRR cohort and n = 10 for PSR cohort, treatment toxicity datas will be reviewed to the IDMC for validation and agreement to continue the study.

OTHER OUTCOMES:
Translational research objectives n°1: Correlation between increase of Tumour Mutational Burden (TMB) after 6 weeks of treatment and response to the treatment combination. | up to 60 months
  TMB will be categorised as high/intermediate/low. TMB after 6 weeks of treatment will be compared to TMB at baseline. Increase is defined as a change in the TMB category.
  Response is defined as clinical and radiological non-progressive disease, as assessed by immune-related response criteria (irRC) (Wolchok et al. 2009) at 3 months in the PRR cohort and 6 months in the PSR cohort.
Translational research objectives n°2: Correlation between Homologous recombination (HR) status at baseline and response to the treatment combination. | up to 60 months
  HR status will be categorised as deficient versus proficient based on genotyping of the baseline biopsy with an HR-genes panel.
  Response is defined as clinical and radiological non-progressive disease, as assessed by immune-related response criteria (irRC) (Wolchok et al. 2009) at 3 months in the PRR cohort and 6 months in the PSR cohort.
Translational research objectives n°3: Correlation between tumour immune infiltrate and Immune Check Point (ICP) status at baseline and response to the association. | up to 60 months
  Immune infiltrate and ICP status of the baseline tumour will be assessed by a targeted transcriptomic approach (IO360 panel, NanoString). Tumours will be categorised as inflamed/excluded/deserted. ICP status will be categorised as "PD-1/PD-L1 driven" versus "others ICPs involved".
  Response is defined as clinical and radiological non-progressive disease, as assessed by immune-related response criteria (irRC) (Wolchok et al. 2009) at 3 months in the PRR cohort and 6 months in the PSR cohort.
  The translational research will provide informations on:
  -Characterization of immune response in the tumor by Nanostring immuno-oncology panel on tumours.

CONTACTS AND LOCATIONS:
Overall Officials: Gilles Freyer, Principal Investigator — Centre Hospitalier Lyon Sud
Locations (9):
- France (9):
  - Institut Bergonié, Bordeaux
  - Centre Oscar Lambret, Lille
  - Centre Léon Bérard, Lyon
  - ICM Val d'Aurelle, Montpellier
  - Groupe Hospitalier des Diaconesses Croix Saint-Simon, Paris
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - Institut Curie - Site Saint Cloud, Saint-Cloud
  - Institut Claudius Régaud, Toulouse
  - Gustave Roussy, Villejuif

IPD SHARING:
Plan to Share IPD: Undecided